CLINICAL TRIAL: NCT05785559
Title: Preliminary Study of Uterine Healing After Caesarean Section: CLInico-ECHOgraphic and Anatomopathologic COrrelation
Acronym: COCLIECHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP220952
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Assessment of Uterine Healing
Keywords: uterine scarring; isthmocele; caesarean section

STUDY DESIGN:
Intervention Model Description: Uterine biopsy and cesarean scar dehiscence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scarred uterus (Experimental): Patients who have already undergone one or more cesarean section(s) during a previous pregnancy and for whom a cesarean section is indicated on a scheduled or emergency basis.
  Interventions: Procedure: uterine biopsies
- Scar dehiscence surgery (Experimental): Patients who have already undergone one or more caesarean section(s) and for whom the surgical management of a dehiscence of a caesarean section scar is indicated outside of pregnancy.
  Interventions: Procedure: uterine biopsies
- Healthy uterus (Experimental): Patients with no history of caesarean section, pregnant with an indication for caesarean section: patients who have never had a caesarean section during a previous pregnancy or who are pregnant with their first pregnancy and for whom a caesarean section is indicated scheduled or urgently"
  Interventions: Procedure: uterine biopsies

INTERVENTIONS:
Procedure: uterine biopsies — uterine biopsies performed on the areas of cesarean section scars

SUMMARY:
Caesarean section is one of the most common surgical procedures. The multiplication of uterine scars leads to an increase in complications and in particular those related to poor healing such as isthmocele or uterine rupture.

The processes of uterine healing at the histological scale are little known. The main objective of the research is to analyze the process of uterine healing by means of uterine biopsies performed on the areas of cesarean section scars.

DETAILED DESCRIPTION:
Our hypothesis is that there is a histological healing defect visible on an anatomopathologic examination of the scar. This poor uterine healing on histological scale is probably associated with uterine healing defects visible on pelvic ultrasound (scar dehiscence) and clinical criteria (number of caesareans, symptoms).

The objective of the research is to analyze uterine scarring by means of uterine biopsies performed on the areas of cesarean section scars. The uterine scarred areas will be analyzed histologically according to specific criteria and compared to healthy uterine areas. Histological characteristics will be compared with clinical and ultrasound data.

ELIGIBILITY:
Inclusion Criteria:

* Common to all groups:
* Adult patient,
* Signed consent for participation in the study
* Patient affiliated to a social security scheme (excluding AME)

Group 1:

* Support for a scheduled or emergency caesarean (excluding patients having an emergency caesarean (red code: caesarean within 15 minutes))
* Scarred uterus: having already benefited from a caesarean section

Group 2:

- Surgical management of caesarean section scar dehiscence after a caesarean section

Group 3 (control):

* Support for a scheduled or emergency caesarean (excluding patients having an emergency caesarean (red code: caesarean within 15 minutes)
* Healthy uterus: no history of caesarean section (history of vaginal delivery or first pregnancy)

Exclusion Criteria:

* Disorder of hemostasis at risk of bleeding
* Anatomopathological sampling not feasible
* Patient with a history of upper genital infections
* Patient under legal protection (guardianship, curatorship)
* Patient who does not speak or understand French
* Patient unable to answer questions or with difficulty in expressing herself

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Analyze the process of uterine healing | 8 weeks
  The main objective of the research is to analyze the process of uterine healing by means of uterine biopsies performed on the areas of cesarean section scars "

SECONDARY OUTCOMES:
Histological aspects of the scar | 8 weeks
  The secondary evaluation criteria will be the correlation of the histological aspects of the scar with the clinical and ultrasound data. The objective is to look for risk factors for poor uterine healing.

CONTACTS AND LOCATIONS:
Overall Officials: Perrine CAPMAS, Principal Investigator — APHP
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No